CLINICAL TRIAL: NCT00983619
Title: A Phase 1, Dose-escalation Study of MEDI-551, a Humanized Monoclonal Antibody Directed Against CD19, in Adult Subjects With Relapsed or Refractory Advanced B-Cell Malignancies
Brief Title: A Clinical Study Using MEDI-551 in Adult Participants With Relapsed or Refractory Advanced B-Cell Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP204; 2009-016378-34 (EudraCT Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: B-cell Malignancies; Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — inebilizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A-MEDI-551 0.5 mg/kg (Experimental): Participants will receive intravenous (IV) infusion of MEDI 551 0.5 mg/kg once every week in 4-week cycles until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part A-MEDI-551 1 mg/kg (Experimental): Participants will receive IV infusion of MEDI 551 1 mg/kg once every week in 4-week cycles until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part A-MEDI-551 2 mg/kg (Experimental): Participants will receive IV infusion of MEDI 551 2 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part A-MEDI-551 4 mg/kg (Experimental): Participants will receive IV infusion of MEDI 551 4 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part A-MEDI-551 8 mg/kg (Experimental): Participants will receive IV infusion of MEDI 551 8 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part A-MEDI-551 12 mg/kg (Experimental): Participants will receive IV infusion of MEDI 551 12 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part B-MEDI-551 6 mg/kg (Experimental): Participants will receive IV infusion of MEDI- 551 6 mg/kg weekly for 4 weeks during Cycle 1 (Days 1, 8, 15, and 22) and thereafter from Cycle 2 on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part B-MEDI-551 12 mg/kg (Experimental): Participants will receive IV infusion of MEDI- 551 12 mg/kg weekly for 4 weeks during Cycle 1 (Days 1, 8, 15, and 22) and thereafter from Cycle 2 on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part B-MEDI-551 24 mg/kg (Experimental): Participants will receive IV infusion of MEDI- 551 24 mg/kg weekly for 4 weeks during Cycle 1 (over 2 days on Day 1 and Day 2, and on Days 8, 15, and 22) and thereafter from Cycle 2, on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
  Interventions: Drug: MEDI-551
- Part C-MEDI-551 8 mg/kg + rituximab (Experimental): Participants will receive IV infusion of MEDI- 551 8 mg/kg on Days 2 and 8 during Cycle 1 and on Day 1 during Cycle 2 (28-day cycle) in combination with rituximab 375 mg/m^2 on Days 1, 8, 15, and 22. From Cycle 3 onwards, only MEDI- 551 8 mg/kg will be administered on Day 1 of each 28-day cycle. The treatment will be continued until the participants experiences unacceptable toxicity, disease progression, reaches complete response or withdraws consent.
  Interventions: Drug: MEDI-551; Drug: Rituximab
- Part C-MEDI-551 12 mg/kg + rituximab (Experimental): Participants will receive IV infusion of MEDI- 551 12 mg/kg on Days 2 and 8 during Cycle 1 and on Day 1 during Cycle 2 (28-day cycle) in combination with rituximab 375 mg/m^2 on Days 1, 8, 15, and 22. From Cycle 3 onwards, only MEDI- 551 8 mg/kg will be administered on Day 1 of each 28-day cycle. The treatment will be continued until the participants experiences unacceptable toxicity, disease progression, reaches complete response or withdraws consent.
  Interventions: Drug: MEDI-551; Drug: Rituximab
- Part D-MEDI-551 12 mg/kg (Experimental): Participants will receive IV infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and thereafter Day 1 of 28- day cycles from Cycle 2 onwards. Treatment will be continued until the participants experiences unacceptable toxicity, disease progression, reaches CR or withdraws consent.
  Interventions: Drug: MEDI-551

INTERVENTIONS:
Drug: MEDI-551 — MEDI-551 will be administered intravenously (IV) once every week in 4-week cycles until complete response, disease progression, toxicity, or another reason for treatment discontinuation will be observed.
Drug: Rituximab — Rituximab will be administered IV on Days 1, 8, 15, and 22 (28- day cycle). The treatment will be continued until the participants experiences unacceptable toxicity, disease progression, reaches complete response or withdraws consent.
  Arms: Part C-MEDI-551 12 mg/kg + rituximab; Part C-MEDI-551 8 mg/kg + rituximab

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of this drug (MEDI-551) in participants with advanced B-cell malignancies. Expansion to occur at maximum tolerated dose (MTD), or if not reached, at optimal biologic dose (OBD).

DETAILED DESCRIPTION:
To determine the MTD or OBD of MEDI-551 in participants with relapsed or refractory advanced B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CLL, DLBCL, FL, or MM;
* Karnofsky Performance Status >= 70;
* Life expectancy of >= 12 weeks;
* Prior radiation therapy provided exposure does not exceed an area of 25% of marrow space
* Adequate hematological function
* Adequate organ function

Exclusion Criteria:

* Any available standard line of therapy known to be life-prolonging or life-saving;
* No concurrent therapy or therapy within six weeks of first dose of MEDI-551 for treatment of cancer
* Previous therapy directed against CD19
* Vaccination (other than experimental cancer vaccine therapy) within 28 days prior to receiving the first dose of MEDI-551;
* History of other invasive malignancy within 5 years except for cervical carcinoma in situ (CIS), non-melanomatous carcinoma of the skin or ductal carcinoma in situ (DCIS) of the breast that have been surgically cured;
* Active infection requiring treatment
* Autologous stem cell transplantation within 4 months prior to study entry;
* Allogeneic stem cell transplantation or any other organ transplant;
* Ongoing >= Grade 2 toxicities from previous cancer therapies unless specifically allowed in the Inclusion/Exclusion criteria.
* Use of immunosuppressive medication other than steroids within 28 days before the first dose of MEDI-551;
* Use of immunosuppressive medication other than steroids within 28 days before the first dose of MEDI-551 (inhaled and topical corticosteroids are permitted);
* Documented current central nervous system involvement by leukemia or lymphoma;
* Pregnancy or lactation;
* Clinically significant abnormality on ECG.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-04-16 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune Inc. Clinical Development, Study Director — MedImmune LLC
Locations (20):
- United States (13):
  - Research Site, Birmingham, Alabama
  - Research Site, La Jolla, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Westwood, Kansas
  - Research Site, Rochester, Minnesota
  - Research Site, New Brunswick, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, Hershey, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Belgium (3):
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Yvoir
- Research Site, Montreal, Quebec, Canada
- Italy (2):
  - Research Site, Cona
  - Research Site, Modena
- Research Site, Madrid, Spain

REFERENCES:
- See also: Click here and search for drug information provided by the FDA. — https://www.fda.gov/safety/medwatch-fda-safety-information-and-adverse-event-reporting-program
- See also: Click here to find results for studies related to marketed products. — https://www.clinicaltrials.gov/
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=MI-CP204&attachmentIdentifier=316ce04f-0e5f-406f-b2be-42b8ce6ae595&fileName=CP204_SAP_v4_Final_Redacted.pdf&versionIdentifier=
- See also: MI-CP204 redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=MI-CP204&attachmentIdentifier=e262f497-135c-41f5-829e-6723fdd242de&fileName=study-protocol-mi-cp204-v13_final_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 137 participants were screened, out of which 1 participant never received the study treatment. A total of 136 participants received study treatment.
Groups:
- Part A-MEDI-551 0.5 mg/kg: Participants received intravenous (IV) infusion of MEDI 551 0.5 mg/kg once every week in 4-week cycles until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part A-MEDI-551 1 mg/kg: Participants received IV infusion of MEDI 551 1 mg/kg once every week in 4-week cycles until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part A-MEDI-551 2 mg/kg: Participants received IV infusion of MEDI 551 2 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part A-MEDI-551 4 mg/kg: Participants received IV infusion of MEDI 551 4 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part A-MEDI-551 8 mg/kg: Participants received IV infusion of MEDI 551 8 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part A-MEDI-551 12 mg/kg: Participants received IV infusion of MEDI 551 12 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part B-MEDI-551 6 mg/kg: Participants received IV infusion of MEDI- 551 6 mg/kg weekly for 4 weeks during Cycle 1 (Days 1, 8, 15, and 22) and thereafter from Cycle 2 on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part B-MEDI-551 12 mg/kg: Participants received IV infusion of MEDI- 551 12 mg/kg weekly for 4 weeks during Cycle 1 (Days 1, 8, 15, and 22) and thereafter from Cycle 2 on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part B-MEDI-551 24 mg/kg: Participants received IV infusion of MEDI- 551 24 mg/kg weekly for 4 weeks during Cycle 1 (over 2 days on Day 1 and Day 2, and on Days 8, 15, and 22) and thereafter from Cycle 2, on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
- Part C-MEDI-551 8 mg/kg + Rituximab: Participants received IV infusion of MEDI- 551 8 mg/kg on Days 2 and 8 during Cycle 1 and on Day 1 during Cycle 2 (28-day cycle) in combination with rituximab 375 mg/m^2 on Days 1, 8, 15, and 22. From Cycle 3 onwards, only MEDI- 551 8 mg/kg was administered on Day 1 of each 28-day cycle. The treatment was continued until the participants experienced unacceptable toxicity, disease progression, reached complete response or withdrew consent.
- Part C-MEDI-551 12 mg/kg + Rituximab: Participants received IV infusion of MEDI- 551 12 mg/kg on Days 2 and 8 during Cycle 1 and on Day 1 during Cycle 2 (28-day cycle) in combination with rituximab 375 mg/m^2 on Days 1, 8, 15, and 22. From Cycle 3 onwards, only MEDI- 551 8 mg/kg was administered on Day 1 of each 28-day cycle. The treatment was continued until the participants experienced unacceptable toxicity, disease progression, reached complete response or withdrew consent.
- Part D-MEDI-551 12 mg/kg: Participants received IV infusion of MEDI-551 12 mg/kg on Days 1 and 8 of Cycle 1 and thereafter Day 1 of 28- day cycles from Cycle 2 onwards. Treatment was continued until the participants experienced unacceptable toxicity, disease progression, reached CR or withdrew consent.
Period: Overall Study
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Started | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17 | 14
Completed | 0 | 0 | 0 | 1 | 0 | 9 | 0 | 1 | 0 | 0 | 6 | 3
Not Completed | 3 | 4 | 3 | 5 | 3 | 67 | 3 | 2 | 1 | 3 | 11 | 11
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 3 | 1 | 23 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 2 | 2 | 1 | 2 | 30 | 1 | 0 | 1 | 2 | 9 | 8
Not completed — Other | 1 | 0 | 0 | 1 | 0 | 12 | 2 | 2 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any treatment of MEDI-551.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg | TOTAL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17 | 14 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (19.5) | 69.5 (12.5) | 64.7 (18.3) | 63.8 (12.7) | 60.0 (12.1) | 64.4 (11.2) | 61.3 (20.8) | 70.0 (7.0) | 78.0 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 68.0 (11.8) | 69.4 (10.8) | 67.9 (11.0) | 65.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 2 | 1 | 30 | 1 | 1 | 1 | 1 | 10 | 5 | 55
  Male | 1 | 4 | 2 | 4 | 2 | 46 | 2 | 2 | 0 | 2 | 7 | 9 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 3 | 4 | 3 | 6 | 3 | 70 | 3 | 3 | 1 | 3 | 17 | 14 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 8
  White | 3 | 3 | 3 | 5 | 3 | 68 | 3 | 2 | 1 | 2 | 15 | 14 | 122
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Optimal Biologic Dose of MEDI-551 for Part A
Description: Optimal biologic dose (OBD) was defined as the dose lower than the maximum tolerated dose (MTD), used for dose expansion. The MTD is defined as the highest dose at which less than equal to (<=) 1 out of 6 participants experience a dose limiting toxicities (DLT) from the time of first administration of MEDI-551 through the first 28-day cycle.
Time Frame: Day 1 to Day 28 of Cycle 1
Population: Dose limiting toxicity evaluable population included all participants in the dose-escalation phase who received at least 1 full cycle of MEDI-551 and completed safety follow-up through the DLT evaluable period (from the time of first administration of MEDI-551 through the first 28-day of cycle 1).
Measure: Number; unit: mg/Kg
Groups:
- Part A-MEDI-551 Part A: Participants received IV infusion of MEDI 551 0.5 or 1 mg/kg (both, once every week in 4-week cycles), or 2, or 4, or 8, or 12 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
Arm/Group | Part A-MEDI-551 Part A
Number analyzed (Participants) | 95
mg/Kg | 12

2. Primary Outcome: Highest Protocol-defined Dose for Part B
Description: Highest protocol-defined dose is dose of MEDI-551 in the absence of exceeding the MTD in participants with relapsed or rituximab-refractory chronic lymphocytic leukemia (defined as those with less than a partial response (PR) or progression within 6 months after completing therapy with rituximab). The MTD is defined as the highest dose at which <= 1 out of 6 participants experience a DLT from the time of first administration of MEDI-551 through the first 28-day cycle.
Time Frame: Day 1 to Day 28 of Cycle 1
Population: DLT evaluable population included all participants in the dose-escalation phase who received at least 1 full cycle of MEDI-551 and completed safety follow-up through the DLT evaluable period (from the time of first administration of MEDI-551 through the first 28-day of cycle).
Measure: Number; unit: mg/Kg
Groups:
- Part B-MEDI-551: Participants received IV infusion of MEDI- 551 6 or 12 mg/kg weekly for 4 weeks during Cycle 1 (both from Days 1, 8, 15, and 22) or 24 mg/kg weekly for 4 weeks during Cycle 1 (over 2 days on Day 1 and Day 2, and on Days 8, 15, and 22) and thereafter from Cycle 2 on Day 1 of each 28-day cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
Arm/Group | Part B-MEDI-551
Number analyzed (Participants) | 7
mg/Kg | 24

3. Primary Outcome: Highest Protocol-defined Dose for Part C
Description: Highest protocol-defined dose is the dose of MEDI-551 in combination with rituximab at the MTD or the highest protocol-defined dose in the absence of exceeding the MTD in participants with aggressive lymphomas. The MTD is defined as the highest dose at which <= 1 out of 6 participants experience a DLT from the time of first administration of MEDI-551 through the first 28-day cycle.
Time Frame: Day 1 to Day 28 of Cycle 1
Population: DLT evaluable population included all participants in the dose-escalation phase who received at least 1 full cycle of MEDI-551 and completed safety follow-up through the DLT evaluable period (from the time of first administration of MEDI-551 through the first 28-day of cycle 1).
Measure: Number; unit: mg/kg
Groups:
- Part C-MEDI-551 + Rituximab: Participants received IV infusion of MEDI- 551 8 or 12 mg/kg on days 2 and 8 during Cycle 1 and on Day 1 during Cycle 2 (28-day cycle) in combination with rituximab 375 mg/m^2 on Days 1, 8, 15, and 22. From Cycle 3 onwards, only MEDI- 551 8 or 12 mg/kg was administered on Day 1 of each 28-day cycle. The treatment was continued until the participants experienced unacceptable toxicity, disease progression, reached complete response or withdraws consent.
Arm/Group | Part C-MEDI-551 + Rituximab
Number analyzed (Participants) | 20
mg/kg | 12

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) for Part A, Part B, and Part C
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17
Participants
  TEAEs | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17
  TESAEs | 1 | 1 | 2 | 1 | 1 | 23 | 1 | 2 | 1 | 1 | 9

5. Primary Outcome: Number of Participants With Dose Limiting Toxicities of MEDI-551 in Part A, Part B, and Part C
Description: A dose limiting toxicities (DLT) for arm A, B, and C was defined as MEDI-551 (or rituximab for Arm C) treatment-related AE of any toxicity grade that led to an inability to receive a full cycle of MEDI-551 (or rituximab for Arm C) or any Grade 3 or higher toxicity (except Grade 3 fever, transient Grade 3 rigors or chills, Grade 3 tumor lysis syndrome, any Grade 3 or 4 electrolyte alteration, any Grade 3 liver function test elevation,>= Grade 3 or 4 lymphopenia or leukopenia, <= Grade 4 neutropenia, <= Grade 4 thrombocytopenia, <= Grade 4 anemia, and Grade 3 infusion-related reaction and infusion reaction), during DLT evaluable period.
Time Frame: Day 1 to Day 28 of Cycle 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs in Part A, Part B, and Part C
Description: Number of participants with clinical laboratory abnormalities reported as TEAEs are reported. Clinical laboratory abnormalities are defined as any abnormal findings in analysis of serum chemistry, hematology, and urine.
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17
Participants
  Anemia | 0 | 2 | 0 | 0 | 1 | 6 | 0 | 1 | 1 | 0 | 4
  Blood fibrinogen decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood fibrinogen increased | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Febrile neutropenia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
  Hematocrit decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Myelocytosis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Neutropenia | 0 | 0 | 0 | 1 | 1 | 14 | 1 | 1 | 0 | 1 | 2
  Neutrophil count abnormal | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 1 | 1 | 0 | 1 | 0 | 5 | 0 | 1 | 1 | 0 | 2
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1
  Red blood cell count decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytosis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Thrombocytopenia | 0 | 1 | 0 | 3 | 0 | 6 | 0 | 1 | 0 | 0 | 2
  White blood cell count decreased | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 2
  Hypergammaglobulinemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Activated PTT prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Blood chloride decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood creatinine increased | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2
  Blood glucose decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood glucose increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood lactate dehydrogenase increased | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
  Blood potassium decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood urea increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood uric acid increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gamma-glutamyl transferase increased | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Hyperbilirubinemia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypercalcemia | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1
  Hyperglycemia | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Hyperkalemia | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperuricemia | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
  Hypocalcemia | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Hypoglycemia | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Hypokalemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Hypomagnesemia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
  Hyponatremia | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Protein total decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood albumin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Hypoalbuminemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Haematuria | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Dysuria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Pollakiuria | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobinuria | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hydronephrosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Urinary incontinence | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in Part A, Part B, and Part C
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal findings in the vital signs parameters (temperature, blood pressure, pulse rate, respiratory rate, and pulse oximetry).
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17
Participants
  Bradycardia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 1
  Dyspnea | 0 | 1 | 1 | 1 | 0 | 10 | 0 | 2 | 1 | 0 | 4
  Hypertension | 2 | 1 | 0 | 0 | 0 | 8 | 0 | 2 | 0 | 0 | 2
  Hypotension | 1 | 3 | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 2
  Orthostatic hypotension | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Palpitations | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Pyrexia | 0 | 0 | 1 | 2 | 0 | 16 | 1 | 1 | 0 | 0 | 3
  Systolic hypertension | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 1

8. Primary Outcome: Number of Participants With Abnormal Electrocardiograms Reported as TEAEs in Part A, Part B, and Part C
Description: Number of participants with abnormal electrocardiograms (ECGs) reported as TEAEs are reported. Abnormal ECGs are defined as any abnormal findings in heart rate, RR interval, PR interval, QRS, axis, and QT intervals from the primary lead of the digital 12-lead ECG.
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 1 | 3 | 17
Participants
  Sinus bradycardia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Atrial fibrillation | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
  Mitral valve incompetence | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Supraventricular extrasystoles | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Tricuspid valve incompetence | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ECG QT prolonged | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Atrial flutter | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Atrial tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Supraventricular tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

9. Primary Outcome: Percentage of Participants With Complete Response for Part B, Part C, and Part D
Description: Complete response (CR) is defined as disappearance of all evidence of disease according to International Working Group criteria (IWG). For nodal masses; fluorodeoxyglucose (FDG)-avid or polyethylene terephthalate (PET) positive prior to therapy; mass of any size permitted if PET negative .Variably FDG-avid or PET negative; regression to normal size on computed tomography (CT). For spleen; not palpable, nodules disappeared. For bone marrow; infiltrate cleared on repeat biopsy; if indeterminate by morphology, immunohistochemistry (IHC) was negative.
Time Frame: Day 1 of all Cycles, then every 2 months during the first year of treatment and then every 6 months until end of treatment (unacceptable toxicity, disease progression, withdraws consent, whichever occurred first) (approximately 9 years)
Population: Evaluable population for efficacy included all participants who received any treatment of MEDI-551 and completed at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 16 | 13
Percentage of Participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8] |  | 33.3 [0.8 to 90.6] | 18.8 [4.0 to 45.6] | 0 [0.0 to 24.7]

10. Primary Outcome: Percentage of Participants With Partial Response for Part B, Part C, and Part D
Description: The PR is defined as regression of measurable disease and no new sites according to IWG criteria. Nodal masses: >= 50% decrease in sum of the product diameters (SPD) of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) FDG-avid or PET negative; regression on CT. Spleen and liver: >= 50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen. Bone marrow: irrelevant if positive prior to therapy.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 16 | 13
Percentage of Participants | 33.3 | 33.3 |  | 33.3 | 25.0 | 23.1

11. Primary Outcome: Duration of Complete Response for Part B, Part C, and Part D
Description: Duration of CR is from the first documentation of a CR to the time of progressive disease/relapse according to IWG criteria. The CR is disappearance of all evidence of disease according to IWG criteria. For nodal masses; FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative. Variably FDG-avid or PET negative; regression to normal size on CT. For spleen; not palpable, nodules disappeared. For bone marrow; infiltrate cleared on repeat biopsy; if indeterminate by morphology, IHC was negative. Kaplan-Meier method was used to evaluate duration of CR.
Time Frame: as for outcome 9
Population: Evaluable population for efficacy included all participants who received any treatment of MEDI-551 and completed at least one post-baseline disease assessment. Duration of CR is calculated for participants with CR.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 3 | 0
Months | NA [5.6 to 5.6] — Median was not estimable because insufficient number of participants had the events. |  |  | NA [0.3 to 0.3] — Median was not estimable because insufficient number of participants had the events. | NA [20.0 to 38.4] — Median was not estimable because insufficient number of participants had the events. |

12. Primary Outcome: Percentage of Participants With Objective Response Rate for Part B, Part C, and Part D
Description: Objective response rate (ORR) is proportion of participants with CR or partial response (PR) as per IWG criteria. CR is disappearance of all evidence of disease. Nodal masses; FDG-avid/PET positive prior to therapy; mass of any size permitted if PET negative. FDG-avid or PET negative; regression to normal size on CT. Spleen; not palpable, nodules disappeared. Bone marrow; infiltrate cleared on repeat biopsy; if unknown by morphology, IHC was negative. PR is regression of measurable disease and no new sites. Nodal masses: >= 50% decrease in sum of the product diameters (SPD) of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) FDG-avid or PET negative; regression on CT. Spleen and liver: >= 50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen. Bone marrow: irrelevant if positive prior to therapy.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 16 | 13
Percentage of participants | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] |  | 66.7 [9.4 to 99.2] | 43.8 [19.8 to 70.1] | 23.1 [5.0 to 53.8]

13. Primary Outcome: Duration of Objective Response for Part B, Part C, and Part D
Description: Duration of objective response (DOR) is the first documentation of objective response to the first documented progressive disease (PD) or relapse according to IWG criteria. PD is defined as any new lesion or increase by >=50% of previously involved sites from nadir. For nodal masses: appearance of a new lesion(s) > 1.5 cm in any axis, >= 50% increase in SPD of more than one node, or >= 50% increase in longest diameter of a previously identified node > 1 cm in short axis lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy. For spleen: > 50% increase from nadir in the SPD of any previous lesions. For bone marrow: New or recurrent involvement. Kaplan-Meier method was used to evaluate DOR.
Time Frame: Cycle 1 Day 1, then every 2 months during the first year of treatment and then every 6 months until end of treatment (unacceptable toxicity, disease progression, withdraws consent, whichever occurred first) (approximately 9 years)
Population: Evaluable population for efficacy included all participants who received any treatment of MEDI-551 and completed at least one post-baseline disease assessment. The DOR were calculated for participants with objective response.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2 | 7 | 3
Months | NA [38.9 to 47.2] — Median was not estimable because insufficient number of participants had the events. | 27.5 [27.5 to 27.5] |  | 3.7 [2.4 to 3.7] | NA [1.0 to 44.7] — Median was not estimable because insufficient number of participants had the events. | 3.7 [1.9 to 27.2]

14. Primary Outcome: Percentage of Participants With Disease Control Rate for Part B, Part C, and Part D
Description: Disease control includes CR, PR, or stable disease (SD) for at least 8 weeks according to IWG criteria. The CR is disappearance of all evidence of disease. Nodal masses; FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative. FDG-avid or PET negative; regression to normal size on CT. Spleen; not palpable, nodules disappeared. Bone marrow; infiltrate cleared on repeat biopsy; if indeterminate by morphology, IHC was negative. PR is regression of measurable disease and no new sites. Nodal masses: >= 50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT. Spleen and liver: >= 50% decrease in SPD of nodules; no increase in size of liver or spleen. For bone marrow: irrelevant if positive prior to therapy. SD is failure to attain CR/PR or PD.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 11 | 6
Percentage of participants | 100 [29.2 to 100] | 100 [29.2 to 100] |  | 100 [29.2 to 100] | 68.8 [41.3 to 89.0] | 46.2 [19.2 to 74.9]

15. Primary Outcome: Duration of Disease Control for Part B, Part C, and Part D
Description: Duration of disease control is defined as the time period from start of MEDI-551 administration to the event of PD/relapse. PD is defined as any new lesion or increase by >=50% of previously involved sites from nadir. For nodal masses: appearance of a new lesion(s) > 1.5 cm in any axis, >= 50% increase in SPD of more than one node, or >= 50% increase in longest diameter of a previously identified node > 1 cm in short axis lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy. For spleen: > 50% increase from nadir in the SPD of any previous lesions. For bone marrow: New or recurrent involvement. Kaplan-Meier method was used to evaluate duration of disease control.
Time Frame: as for outcome 9
Population: Evaluable population for efficacy included all participants who received any treatment of MEDI-551 and completed at least one post-baseline disease assessment. Duration of disease control is calculated for the participants with objective response or stable disease response.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 11 | 6
Months | NA [9.7 to 50.9] — Median was not estimable because insufficient number of participants had the events. | 29.8 [22.6 to 39.5] |  | 5.5 [4.2 to 5.5] | 14.6 [1.7 to 46.5] | 3.8 [3.5 to 29.0]

16. Primary Outcome: Time to Response for Part B, Part C, and Part D
Description: Time to response (TTR) is measured from the start of MEDI-551 administration to the first documentation of response (CR or PR) and assessed in participants who have achieved objective response. Kaplan-Meier method was used to evaluate TTR.
Time Frame: as for outcome 9
Population: Evaluable population for efficacy included all participants who received any treatment of MEDI-551 and completed at least one post-baseline disease assessment. TTR were calculated for the participants with objective response.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 2 | 1 | 0 | 2 | 7 | 3
Months | 6.5 [3.7 to 9.2] | 12.0 [12.0 to 12.0] |  | 1.8 [1.7 to 1.8] | 2.0 [1.7 to 17.3] | 1.8 [1.6 to 1.9]

17. Primary Outcome: Progression Free Survival for Part B, Part C, and Part D
Description: Progression-free survival (PFS) is measured from the start of MEDI-551 treatment until the first documentation of disease progression, relapse or death, whichever occurs first. The PFS was censored on the date of last disease assessment for participants who have no documented PD/relapse or death prior to data cutoff, dropout, or the initiation of alternative anticancer therapy. Kaplan-Meier method was used to evaluate PFS.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 16 | 13
Months | NA [9.7 to 50.9] — Median was not estimable because insufficient number of participants had the events. | 29.8 [22.6 to 39.5] |  | 5.5 [4.2 to 5.5] | 3.5 [0.7 to 46.5] | 2.0 [0.7 to 29.0]

18. Primary Outcome: Overall Survival for Part B, Part C, and Part D
Description: Overall survival (OS) is measured from the start of MEDI-551 treatment until death. For participants who are alive at the end of study or lost to follow-up, OS will be censored on the last date when participants were known to be alive. Kaplan-Meier method was used to evaluate OS.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 3 | 0 | 3 | 16 | 13
Months | NA [19.4 to 53.8] — Median was not estimable because insufficient number of participants had the events. | NA [37.6 to 41.9] — Median was not estimable because insufficient number of participants had the events. |  | 25.0 [18.3 to 45.4] | 33.4 [0.9 to 51.3] | 17.9 [1.2 to 38.9]

19. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) for Part D
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 14
Participants
  TEAEs | 14
  TESAEs | 5

20. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs in Part D
Description: as for outcome 6
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 14
Participants
  Anemia | 2
  Febrile neutropenia | 1
  Lymphocyte count decreased | 3
  Neutropenia | 1
  Neutrophil count decreased | 4
  Platelet count decreased | 1
  Polycythemia | 1
  Thrombocytopenia | 2
  White blood cell count decreased | 3
  Blood ALP increased | 1
  Blood bilirubin increased | 1
  Blood LDH increased | 1
  Blood potassium decreased | 1
  Hypercalcemia | 1
  Hyperglycemia | 2
  Hyperuricemia | 2
  Hypocalcemia | 1
  Hypokalemia | 2
  Pollakiuria | 1
  Urinary incontinence | 1

21. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in Part D
Description: as for outcome 7
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 14
Participants
  Chills | 2
  Dyspnea | 1
  Hypertension | 1
  Hypotension | 1
  Palpitations | 1
  Pyrexia | 2
  Tachycardia | 1

22. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms Reported as TEAEs in Part D
Description: Number of participants with abnormal ECGs reported as TEAEs are reported. Abnormal ECGs are defined as any abnormal findings in heart rate, RR interval, PR interval, QRS, axis, and QT intervals from the primary lead of the digital 12-lead ECG.
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Count of Participants; unit: Participants
Arm/Group | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 14
Participants | 1

23. Secondary Outcome: Percentage of Participants With Complete Response for Part A
Description: The CR is defined as disappearance of all evidence of disease according to IWG criteria. For nodal masses; FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative .Variably FDG-avid or PET negative; regression to normal size on CT. For spleen; not palpable, nodules disappeared. For bone marrow; infiltrate cleared on repeat biopsy; if indeterminate by morphology, IHC was negative.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 72
Percentage of Participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 20.0 [0.5 to 71.6] | 0 [0.0 to 70.8] | 12.5 [5.9 to 22.4]

24. Secondary Outcome: Percentage of Participants With Partial Response for Part A
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 72
Percentage of Participants | 33.3 | 0 | 0 | 0 | 33.3 | 15.3

25. Secondary Outcome: Duration of Complete Response for Part A
Description: Duration of CR is from the first documentation of a CR to the time of progressive disease/relapse according to IWG criteria. The CR is disappearance of all evidence of disease. For nodal masses; FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative. Variably FDG-avid or PET negative; regression to normal size on CT. For spleen; not palpable, nodules disappeared. For bone marrow; infiltrate cleared on repeat biopsy; if indeterminate by morphology, IHC was negative. Kaplan-Meier method was used to evaluate duration of CR.
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Median (Full Range); unit: Months
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 9
Months | 7.1 [7.1 to 7.1] |  |  | 14.9 [14.9 to 14.9] |  | 14.3 [1.9 to 31.8]

26. Secondary Outcome: Percentage of Participants With Objective Response Rate for Part A
Description: The ORR is defined as proportion of participants with CR or PR according to IWG criteria. CR is disappearance of all evidence of disease. For nodal masses; FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative. FDG-avid or PET negative; regression to normal size on CT. For spleen; not palpable, nodules disappeared. For bone marrow; infiltrate cleared on repeat biopsy; if unknown by morphology, IHC was negative. PR is regression of measurable disease and no new sites. For nodal masses: >= 50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) FDG-avid or PET negative; regression on CT. For spleen and liver: >= 50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen. For bone marrow: irrelevant if positive prior to therapy.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 72
Percentage of participants | 66.7 [9.4 to 99.2] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 20.0 [0.5 to 71.6] | 33.3 [0.8 to 90.6] | 27.8 [17.9 to 39.6]

27. Secondary Outcome: Duration of Objective Response for Part A
Description: The DOR is the first documentation of objective response to the first documented PD or relapse according to IWG criteria. PD is defined as any new lesion or increase by >=50% of previously involved sites from nadir. For nodal masses: appearance of a new lesion(s) > 1.5 cm in any axis, >= 50% increase in SPD of more than one node, or >= 50% increase in longest diameter of a previously identified node > 1 cm in short axis lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy. For spleen: > 50% increase from nadir in the SPD of any previous lesions. For bone marrow: New or recurrent involvement. Kaplan-Meier method was used to evaluate DOR.
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Median (Full Range); unit: Months
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 2 | 0 | 0 | 1 | 1 | 20
Months | 8.8 [7.4 to 8.8] |  |  | 15.0 [15.0 to 15.0] | 3.0 [3.0 to 3.0] | 19.8 [0.0 to 41.9]

28. Secondary Outcome: Percentage of Participants With Disease Control Rate for Part A
Description: Disease control includes CR, PR, or SD for at least 8 weeks according to IWG criteria. The CR is disappearance of all evidence of disease. For nodal masses; FDG -avid or PET positive prior to therapy; mass of any size permitted if PET negative. FDG-avid or PET negative; regression to normal size on CT. For spleen; not palpable, nodules disappeared. For bone marrow; infiltrate cleared on repeat biopsy; if indeterminate by morphology, IHC was negative. PR is regression of measurable disease and no new sites. For nodal masses: >= 50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT. For spleen and liver: >= 50% decrease in SPD of nodules; no increase in size of liver or spleen. For bone marrow: irrelevant if positive prior to therapy. SD is failure to attain CR/PR or PD.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 72
Percentage of participants | 66.7 [9.4 to 99.2] | 50.0 [6.8 to 93.2] | 66.7 [9.4 to 99.2] | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2] | 73.6 [61.9 to 83.3]

29. Secondary Outcome: Duration of Disease Control for Part A
Description: Duration of disease control is defined as the time period from start of MEDI-551 administration to the event of PD/relapse according to IWG criteria. PD is defined as any new lesion or increase by >=50% of previously involved sites from nadir. For nodal masses: appearance of a new lesion(s) > 1.5 cm in any axis, >= 50% increase in SPD of more than one node, or >= 50% increase in longest diameter of a previously identified node > 1 cm in short axis lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy. For spleen: > 50% increase from nadir in the SPD of any previous lesions. For bone marrow: New or recurrent involvement. Kaplan-Meier method was used to evaluate duration of disease control.
Time Frame: as for outcome 9
Population: as for outcome 15
Measure: Median (Full Range); unit: Months
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 2 | 53
Months | 12.6 [1.4 to 12.6] | NA [9.4 to 21.0] — Median was not estimable because insufficient number of participants had the events. | NA [3.5 to 7.4] — Median was not estimable because insufficient number of participants had the events. | 10.9 [3.9 to 94.9] | 6.6 [2.8 to 6.6] | 18.0 [0.9 to 49.7]

30. Secondary Outcome: Time to Response for Part A
Description: The TTR is measured from the start of MEDI-551 administration to the first documentation of response (CR or PR) and assessed in participants who have achieved objective response. Kaplan-Meier method was used to evaluate TTR.
Time Frame: as for outcome 9
Population: as for outcome 16
Measure: Median (Full Range); unit: Months
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 2 | 0 | 0 | 1 | 1 | 20
Months | 3.7 [3.5 to 3.9] |  |  | 1.9 [1.9 to 1.9] | 3.6 [3.6 to 3.6] | 3.2 [0.3 to 22.6]

31. Secondary Outcome: Progression Free Survival for Part A
Description: The PFS is measured from the start of MEDI-551 treatment until the first documentation of disease progression, relapse or death, whichever occurs first. Kaplan-Meier method was used to evaluate PFS. The PFS was censored on the date of last disease assessment for participants who have no documented PD/relapse or death prior to data cutoff, dropout, or the initiation of alternative anticancer therapy.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 72
Months | 12.6 [1.4 to 12.6] | 5.9 [0.6 to 21.0] | 3.5 [1.6 to 9.9] | 4.9 [1.1 to 94.9] | 6.6 [2.1 to 6.6] | 11.3 [0.0 to 49.7]

32. Secondary Outcome: Overall Survival for Part A
Description: The OS is measured from the start of MEDI-551 treatment until death. For participants who are alive at the end of study or lost to follow-up, OS will be censored on the last date when participants were known to be alive. Kaplan-Meier method was used to evaluate OS.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 72
Months | NA [1.4 to 21.5] — Median was not estimable because insufficient number of participants had the events. | 44.6 [0.8 to 91.5] | 9.9 [2.8 to 9.9] | NA [1.7 to 94.9] — Median was not estimable because insufficient number of participants had the events. | 8.1 [2.8 to 12.5] | 45.3 [0.7 to 83.5]

33. Secondary Outcome: Trough Serum Concentration of MEDI-551 by Treatment Cycle
Description: Trough serum concentration (Ctrough) is defined as lowest concentration reached by a drug before the next dose is administered. The Ctrough concentration of MEDI-551 by treatment cycle is reported.
Time Frame: For Part A: C1D1 of each cycles; For Part B: C1D1 of each cycle + C1D8, C1D15, and C1D22; For Part C: C1D2, C1D8, then Day 1 of each cycle until Cycle 10;For Part D: C1D1, C1D8, then Day 1 of each cycle until Cycle 10
Population: Pharmacokinetic population included all participants who received at least one dose of MEDI-551 and had at least one measurable serum concentration of MEDI-551. The "Number of Participants Analyzed" denotes the number of participants evaluated for specific day.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Part A-MEDI-551 12 mg/kg (Expansion): Participants received IV infusion of MEDI 551 12 mg/kg on Days 1 and 8 of Cycle 1 (loading doses) and then once every 28 days at the start of each subsequent cycle until complete response, disease progression, toxicity, or another reason for treatment discontinuation was observed.
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part A-MEDI-551 12 mg/kg (Expansion) | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 17 | 14
μg/mL
  Cycle 1 (C1) Day 1 (D1): number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 66 | 3 | 3 | 1 | 3 | 17 | 14
  Cycle 1 (C1) Day 1 (D1) | NA (NA) — The sample was below limit of quantification. | 0.333 (0.665) | NA (NA) — The sample was below limit of quantification. | NA (NA) — The sample was below limit of quantification. | NA (NA) — The sample was below limit of quantification. | NA (NA) — The sample was below limit of quantification. | 2.97 (24.1) | NA (NA) — The sample was below limit of quantification. | NA (NA) — The sample was below limit of quantification. | NA (NA) — The sample was below limit of quantification. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — The sample was below limit of quantification.
  C1D2 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — The sample was below limit of quantification. | NA (NA) — The sample was below limit of quantification. | NA (NA) — Not applicable for this arm.
  C1D8: number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 16 | 14
  C1D8 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 46.5 (20.9) | 102 (25.0) | 125 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 58.0 (14.3) | 115 (38.0) | 109 (58.5)
  C1D15 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 81.8 (38.3) | 197 (51.2) | 329 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm.
  C1D22: number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 0 | 3 | 17 | 14
  C1D22 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 116 (47.4) | 281 (29.5) |  | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm.
  C2D1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 6 | 56 | 3 | 3 | 0 | 3 | 12 | 11
  C2D1 | 15.6 (0.823) | 25.9 (10.9) | 12.9 (4.55) | 59.4 (11.0) | 89.8 (64.9) | 166 (54.0) | 124 (64.8) | 122 (37.2) | 326 (68.0) |  | 52.4 (17.7) | 106 (28.8) | 114 (40.1)
  C3D1: number analyzed (Participants) | 2 | 3 | 2 | 4 | 2 | 6 | 46 | 3 | 3 | 0 | 3 | 11 | 6
  C3D1 | 19.3 (3.33) | 26.9 (12.2) | 6.78 (2.01) | 43.0 (8.40) | 97.0 (94.5) | 149 (46.2) | 113 (70.3) | 57.6 (43.1) | 187 (80.6) |  | 44.7 (14.2) | 92.1 (30.7) | 93.9 (35.6)
  C4D1: number analyzed (Participants) | 2 | 2 | 2 | 4 | 1 | 5 | 43 | 3 | 3 | 0 | 3 | 10 | 6
  C4D1 | 20.9 (6.69) | 36.5 (0.550) | 5.59 (0.146) | 37.9 (13.8) | 33.4 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 146 (55.5) | 113 (57.1) | 36.0 (31.6) | 134 (67.7) |  | 48.2 (20.8) | 113 (70.0) | 102 (61.5)
  C5D1: number analyzed (Participants) | 2 | 2 | 0 | 3 | 1 | 3 | 34 | 3 | 3 | 0 | 2 | 7 | 2
  C5D1 | 26.6 (7.17) | 46.8 (8.03) |  | 56.9 (19.6) | 31.8 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 136 (19.3) | 117 (60.9) | 35.7 (32.0) | 121 (78.1) |  | 51.6 (2.64) | 102 (26.3) | 147 (105)
  C6D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 1 | 3 | 35 | 3 | 3 | 0 | 1 | 7 | 2
  C6D1 | 29.1 (6.17) | 29.1 (17.3) | 11.7 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 32.0 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 33.7 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 138 (27.2) | 123 (67.9) | 37.3 (33.5) | 106 (54.6) |  | 45.9 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 100 (22.9) | 150 (116)
  C7D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 1 | 3 | 28 | 3 | 3 | 0 | 1 | 5 | 1
  C7D1 | 31.4 (7.08) | 25.1 (27.8) | 9.93 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 38.2 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 27.9 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 144 (42.4) | 109 (64.2) | 28.1 (21.2) | 95.1 (54.4) |  | 45.3 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 108 (20.2) | 248 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm.
  C8D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 0 | 1 | 27 | 3 | 3 | 0 | 0 | 5 | 1
  C8D1 | 27.1 (14.9) | 28.0 (1.86) | 8.80 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 33.3 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 109 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 114 (63.8) | 30.8 (30.4) | 86.8 (54.4) |  |  | 147 (82.2) | 177 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm.
  C9D1: number analyzed (Participants) | 1 | 2 | 1 | 1 | 0 | 2 | 22 | 3 | 3 | 0 | 0 | 5 | 2
  C9D1 | 21.6 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 31.6 (1.23) | 10.7 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 33.6 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 124 (23.2) | 121 (77.5) | 27.3 (27.1) | 94.8 (69.4) |  |  | 95.0 (7.59) | 192 (25.9)
  C10D1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 2 | 23 | 3 | 3 | 0 | 0 | 4 | 1
  C10D1 | 17.6 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 25.1 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 10.6 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 32.9 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 98.3 (5.05) | 139 (80.4) | 33.4 (34.8) | 84.2 (57.4) |  |  | 113 (27.6) | 215 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm.

34. Secondary Outcome: Peak Serum Concentration of MEDI-551 by Treatment Cycle
Description: Peak serum concentration is concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part A-MEDI-551 12 mg/kg (Expansion) | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 17 | 14
μg/mL
  Cycle 1 (C1) Day 1 (D1): number analyzed (Participants) | 3 | 4 | 3 | 4 | 3 | 6 | 62 | 3 | 3 | 1 | 3 | 17 | 13
  Cycle 1 (C1) Day 1 (D1) | 12.3 (1.20) | 22.8 (1.24) | 46.0 (22.2) | 100 (11.0) | 166 (59.5) | 280 (99.1) | 240 (90.0) | 122 (24.2) | 335 (79.1) | 199 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 260 (87.3)
  C1D2 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 160 (23.5) | 214 (79.9) | NA (NA) — Not applicable for this arm.
  C1D8: number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 16 | 13
  C1D8 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 162 (17.3) | 393 (80.8) | 470 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 246 (76.1) | 115 (38.0) | 303 (97.4)
  C1D15 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 182 (31.1) | 517 (135) | 619 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm.
  C1D22: number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 0 | 3 | 17 | 14
  C1D22 | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | 208 (46.7) | 533 (223) |  | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm. | NA (NA) — Not applicable for this arm.
  C2D1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 3 | 6 | 53 | 3 | 3 | 0 | 3 | 12 | 10
  C2D1 | 27.5 (0.752) | 43.9 (13.2) | 48.8 (21.7) | 149 (29.7) | 238 (106) | 467 (114) | 350 (130) | 186 (116) | 749 (133) |  | 205 (33.5) | 304 (108) | 333 (72.7)
  C3D1: number analyzed (Participants) | 2 | 3 | 2 | 4 | 2 | 6 | 46 | 3 | 3 | 0 | 3 | 11 | 6
  C3D1 | 26.3 (2.20) | 46.4 (16.6) | 58.7 (0.783) | 145 (31.2) | 260 (89.6) | 374 (116) | 326 (110) | 155 (38.2) | 374 (125) |  | 192 (78.1) | 311 (74.0) | 277 (95.7)
  C4D1: number analyzed (Participants) | 2 | 2 | 2 | 4 | 1 | 5 | 41 | 3 | 3 | 0 | 3 | 10 | 6
  C4D1 | 30.3 (5.46) | 48.3 (12.7) | 63.7 (35.1) | 161 (85.6) | 201 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 359 (115) | 342 (119) | 156 (81.7) | 384 (169) |  | 212 (84.1) | 261 (99.4) | 295 (116)
  C5D1: number analyzed (Participants) | 2 | 2 | 0 | 2 | 1 | 3 | 32 | 3 | 3 | 0 | 2 | 7 | 2
  C5D1 | 39.4 (6.85) | 70.8 (5.43) |  | 151 (58.1) | 203 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 372 (113) | 347 (98.1) | 153 (71.6) | 363 (261) |  | 250 (82.3) | 290 (66.0) | 338 (245)
  C6D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 1 | 3 | 35 | 3 | 3 | 0 | 1 | 6 | 2
  C6D1 | 40.4 (3.87) | 34.4 (4.21) | 43.2 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 123 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 198 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 345 (101) | 337 (82.1) | 130 (45.7) | 349 (140) |  | 209 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 332 (102) | 303 (237)
  C7D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 1 | 3 | 27 | 3 | 3 | 0 | 1 | 5 | 1
  C7D1 | 41.3 (4.72) | 39.5 (30.8) | 41.0 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 123 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 182 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 383 (54.6) | 355 (95.7) | 174 (60.4) | 333 (133) |  | 235 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 392 (93.0) | 502 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm.
  C8D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 0 | 1 | 26 | 3 | 3 | 0 | 0 | 5 | 1
  C8D1 | 29.9 (12.3) | 58.2 (16.9) | 32.2 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 130 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 409 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 367 (102) | 164 (52.0) | 342 (173) |  |  | 317 (150) | 511 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm.
  C9D1: number analyzed (Participants) | 1 | 2 | 1 | 1 | 0 | 2 | 22 | 3 | 3 | 0 | 0 | 5 | 2
  C9D1 | 32.2 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 46.8 (5.58) | 37.8 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 127 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 391 (79.6) | 394 (125) | 159 (64.7) | 299 (69.8) |  |  | 363 (90.3) | 593 (200)
  C10D1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 2 | 21 | 3 | 3 | 0 | 0 | 4 | 1
  C10D1 | 43.3 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 33.5 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 42.3 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 133 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 307 (49.8) | 394 (157) | 166 (64.1) | 316 (189) |  |  | 349 (70.4) | 484 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm.

35. Secondary Outcome: Area Under the Concentration Curve at Steady State (AUCss) of MEDI-551
Description: Area under the concentration-time curve at steady state (Css, AUC) of MEDI-551 is reported.
Time Frame: Part A:Cycle(C)1 Day(D)1 (Pre & post dose [PPD] 2,6,24,48 hrs PD); PPD once a week in 4 weeks C till C71; Part B:C1 (D1,D8,D15,D22),PPD of D1 of each C till C28; Part C & D:PPD of C1 (D2,D8), predose D15 and 22, PPD of D1 of each C till C24
Population: Pharmacokinetic population included all participants who received at least one dose of MEDI-551 and had at least one measurable serum concentration of MEDI-551.
Measure: Mean (Standard Deviation); unit: μg⋅day/mL
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part A-MEDI-551 12 mg/kg (Expansion) | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 17 | 14
μg⋅day/mL | 212 (28.1) | 287 (110) | 479 (57.7) | 1660 (778) | 2880 (2190) | 5720 (1620) | 4850 (1720) | 1730 (1030) | 4920 (1440) | NA (NA) — Data not reported due to limited PK data up to Cycle 1 Day 15. | 2240 (338) | 4260 (1340) | 4250 (2000)

36. Secondary Outcome: Apparent Clearance of MEDI-551
Description: Apparent clearance of MEDI-551 is reported.
Time Frame: as for outcome 35
Population: Population pharmacokinetic model included all participants who received at least one dose of MEDI-551 and provided at least one measurable serum concentration of MEDI-551.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part A-MEDI-551 12 mg/kg (Expansion) | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 17 | 14
mL/day | 206 (101) | 302 (173) | 373 (70.9) | 210 (28.9) | 268 (126) | 198 (44.3) | 235 (110) | 303 (108) | 243 (81.6) | 279 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 288 (43.0) | 235 (87.5) | 237 (72.5)

37. Secondary Outcome: Volume of Distribution of MEDI-551
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Central volume of distribution (Vd1) is defined as hypothetical volume into which a drug initially distributes upon administration and peripheral volume of distribution (Vd2) is defined as the sum of all tissue spaces outside the central compartment.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part A-MEDI-551 12 mg/kg (Expansion) | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 17 | 14
mL
  Vd1 | 3970 (851) | 3920 (491) | 4350 (948) | 4070 (464) | 4210 (510) | 4230 (234) | 4450 (889) | 3560 (286) | 4490 (947) | 5690 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 4520 (126) | 4350 (851) | 4510 (647)
  Vd2 | 2670 (351) | 2010 (1080) | 1980 (888) | 2290 (767) | 2620 (1240) | 2920 (1070) | 3430 (2250) | 3290 (1440) | 2640 (1840) | 3670 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 4590 (847) | 2640 (1200) | 3200 (1440)

38. Secondary Outcome: Terminal Half-life (t1/2) of MEDI-551
Description: Terminal half-life is the time required for the plasma concentration of MEDI-551 to fall by 50% during the terminal phase.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part A-MEDI-551 12 mg/kg (Expansion) | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 6 | 67 | 3 | 3 | 1 | 3 | 17 | 14
Days | 26.0 (6.88) | 17.3 (7.65) | 13.3 (6.41) | 22.1 (3.26) | 21.7 (8.65) | 27.9 (9.08) | 28.9 (15.0) | 19.9 (9.34) | 23.8 (10.9) | 25.1 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 25.3 (4.40) | 23.6 (9.38) | 25.6 (7.96)

39. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) Titer to MEDI-551
Description: Number of participants with positive Anti-drug antibodies (ADA) titer to MEDI-551 is reported.
Time Frame: Part A:C1D1; Part B: C1D1; Part C: C1D1; Part D: C1D1; End of treatment (EOT); 90 Days post last dose (approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551. Participants only with positive ADA is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76 | 3 | 3 | 3 | 17 | 14
Participants
  C1D1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  EOT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  90 Day Post Dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: B-cell Concentration in Serum
Description: B-cell Concentration in serum is reported.
Time Frame: Part A:C1D1 of each cycles; Part B: C1D1 of each cycle + C1D8, C1D15, and C1D22; Part C: C1D2, C1D8, then Day 1 of each cycle until Cycle 10; Part D: C1D1, C1D8, Day 1 of each cycle until Cycle 10; EOT;90 Days post last dose (approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551. It was pre-specified that B-cell analysis was not required, due to limited data availability.
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Immunoglobulin (Ig) Concentration in Serum
Description: Immunoglobin (Ig) concentration in serum is reported.
Time Frame: Part A:C1D1 of each cycles; EOT;90 Days post last dose (approximately 9 years)
Population: Safety population included all participants who received any treatment of MEDI-551.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 76
mg/dL
  C1D1: number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 68
  C1D1 | 120.00 (46.36) | 110.00 (76.25) | 81.00 (66.36) | 61.67 (54.52) | 93.33 (46.11) | 93.01 (88.56)
  C2D1: number analyzed (Participants) | 2 | 3 | 3 | 4 | 2 | 59
  C2D1 | 67.50 (7.78) | 113.67 (92.81) | 67.67 (58.05) | 57.00 (47.05) | 74.50 (47.38) | 88.90 (92.05)
  C3D1: number analyzed (Participants) | 2 | 3 | 2 | 4 | 2 | 50
  C3D1 | 62.50 (6.36) | 106.00 (87.93) | 31.00 (29.70) | 57.25 (48.29) | 76.50 (50.20) | 67.90 (66.59)
  C4D1: number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 50
  C4D1 | 64.00 (9.90) | 152.50 (13.44) | 31.00 (33.94) | 63.67 (56.52) | 98.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 66.84 (61.83)
  C5D1: number analyzed (Participants) | 2 | 2 | 1 | 3 | 1 | 38
  C5D1 | 69.00 (11.31) | 145.50 (38.89) | 50.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 58.67 (45.17) | 77.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 69.24 (70.45)
  C6D1: number analyzed (Participants) | 2 | 2 | 0 | 1 | 1 | 36
  C6D1 | 63.50 (13.44) | 156.00 (48.08) |  | 41.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 71.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 62.86 (65.04)
  C7D1: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 31
  C7D1 | 56.00 (1.41) | 127.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 47.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 41.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 61.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 67.26 (69.36)
  C8D1: number analyzed (Participants) | 2 | 2 | 1 | 1 | 0 | 29
  C8D1 | 47.00 (7.07) | 147.00 (28.28) | 45.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 41.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 73.76 (66.87)
  C9D1: number analyzed (Participants) | 1 | 2 | 1 | 1 | 0 | 26
  C9D1 | 51.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 137.50 (30.41) | 46.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 41.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 62.35 (61.90)
  C10D1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 24
  C10D1 | 47.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 155.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 46.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 41.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. |  | 73.17 (66.34)
  EOT: number analyzed (Participants) | 2 | 3 | 3 | 5 | 3 | 48
  EOT | 43.50 (12.02) | 96.00 (80.58) | 7.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 54.40 (46.55) | 65.33 (19.76) | 217.25 (1003.38)
  90 Days Post Dose: number analyzed (Participants) | 1 | 2 | 0 | 3 | 0 | 15
  90 Days Post Dose | 49.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 84.50 (60.10) |  | 93.33 (42.06) |  | 45.20 (38.72)

ADVERSE EVENTS:
Time Frame: Day 1 through 90-Day Post Last Dose (Approximately 9 years)
Arm/Group | Part A-MEDI-551 0.5 mg/kg | Part A-MEDI-551 1 mg/kg | Part A-MEDI-551 2 mg/kg | Part A-MEDI-551 4 mg/kg | Part A-MEDI-551 8 mg/kg | Part A-MEDI-551 12 mg/kg | Part B-MEDI-551 6 mg/kg | Part B-MEDI-551 12 mg/kg | Part B-MEDI-551 24 mg/kg | Part C-MEDI-551 8 mg/kg + Rituximab | Part C-MEDI-551 12 mg/kg + Rituximab | Part D-MEDI-551 12 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/4 | 2/3 | 1/6 | 2/3 | 30/76 | 1/3 | 0/3 | 1/1 | 2/3 | 9/17 | 8/14
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 2/3 | 1/6 | 1/3 | 23/76 | 1/3 | 2/3 | 1/1 | 1/3 | 9/17 | 5/14
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/6 | 3/3 | 75/76 | 3/3 | 3/3 | 1/1 | 3/3 | 17/17 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A-MEDI-551 0.5 mg/kg (N=3) | Part A-MEDI-551 1 mg/kg (N=4) | Part A-MEDI-551 2 mg/kg (N=3) | Part A-MEDI-551 4 mg/kg (N=6) | Part A-MEDI-551 8 mg/kg (N=3) | Part A-MEDI-551 12 mg/kg (N=76) | Part B-MEDI-551 6 mg/kg (N=3) | Part B-MEDI-551 12 mg/kg (N=3) | Part B-MEDI-551 24 mg/kg (N=1) | Part C-MEDI-551 8 mg/kg + Rituximab (N=3) | Part C-MEDI-551 12 mg/kg + Rituximab (N=17) | Part D-MEDI-551 12 mg/kg (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A-MEDI-551 0.5 mg/kg (N=3) | Part A-MEDI-551 1 mg/kg (N=4) | Part A-MEDI-551 2 mg/kg (N=3) | Part A-MEDI-551 4 mg/kg (N=6) | Part A-MEDI-551 8 mg/kg (N=3) | Part A-MEDI-551 12 mg/kg (N=76) | Part B-MEDI-551 6 mg/kg (N=3) | Part B-MEDI-551 12 mg/kg (N=3) | Part B-MEDI-551 24 mg/kg (N=1) | Part C-MEDI-551 8 mg/kg + Rituximab (N=3) | Part C-MEDI-551 12 mg/kg + Rituximab (N=17) | Part D-MEDI-551 12 mg/kg (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 4 (18) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 13 (19) | 1 (1) | 1 (13) | 0 (0) | 1 (1) | 2 (7) | 1 (2)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 0 (0) | 6 (7) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (19) | 2 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 6 (7) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (10) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 18 (21) | 1 (1) | 2 (3) | 1 (2) | 1 (1) | 5 (15) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 13 (16) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 5 (9) | 3 (3)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Breakthrough pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (5) | 1 (1) | 2 (2) | 3 (3) | 28 (33) | 2 (2) | 3 (6) | 0 (0) | 1 (2) | 9 (20) | 5 (6)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Gravitational oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Necrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 2 (5) | 1 (2) | 0 (0) | 5 (9) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 13 (18) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (7) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (6) | 1 (2) | 0 (0) | 0 (0) | 4 (8) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 2 (6) | 1 (10) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 34 (108) | 1 (6) | 2 (8) | 1 (1) | 0 (0) | 1 (1) | 4 (12)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin m decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood triglycerides increased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Karnofsky scale worsened (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 0 (0) | 2 (7) | 3 (3)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (5) | 0 (0) | 1 (4) | 0 (0) | 5 (7) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 2 (4) | 1 (8) | 0 (0) | 2 (4) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 3 (6) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 11 (12) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 4 (5) | 2 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 15 (20) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 4 (4)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 26 (31) | 1 (1) | 3 (7) | 0 (0) | 0 (0) | 3 (3) | 2 (5)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 9 (10) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (19) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ex-tobacco user (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (4) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medimmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT00983619/SAP_000.pdf
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT00983619/Prot_001.pdf